CLINICAL TRIAL: NCT00475813
Title: Study of FLUTIFORM® VS Seretide® in Paediatric Subjects With Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mundipharma Research Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: FLT3502; 2006-005928-16
Record Dates: First submitted 2007-05-18; First posted 2007-05-21 (Estimated); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Asthma
Keywords: Paediatric subjects with asthma
MeSH Terms: conditions — Asthma | interventions — fluticasone-formoterol; Formoterol Fumarate; Fluticasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: FLUTIFORM® (Formoterol fumarate / Fluticasone propionate)

SUMMARY:
Study compares the efficacy and safety of FLUTIFORM® with Seretide® in the treatment of mild to moderate persistent asthma in pediatric subjects.

DETAILED DESCRIPTION:
This is a study involving a 12 week treatment phase followed by a 6 month extension phase. During the treatment phase subjects receive FLUTIFORM® or Seretide®. In the extension phase all subjects receive FLUTIFORM®. Efficacy will be assessed by lung function tests and asthma symptoms, sleep disturbance. Safety will be assessed by adverse events, vital signs, lab tests and ECGs.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients between 4-12 years of age. Female patients must be pre-menarche to be eligible.
* Known history of mild to moderate reversible asthma for ≥ 6 months prior to the screening visit.
* Demonstrate a FEV1 of ≥60% to ≤80% of predicted normal values (Zapletal, 1977) during the screening phase following appropriate withholding of asthma medications (if applicable).

  * No beta agonist use on day of screening.
  * No use of combination asthma therapy on day of screening.
  * Inhaled corticosteroids are allowed on day of screening.
* Documented reversibility of ≥ 15% in FEV1 during the screening phase.
* Demonstrate satisfactory technique in the use of the pressurized MDI and spacer device.
* Willing and able to enter information in the electronic diary (parental help is acceptable for young children) and attend all study visits.
* Willing and able to substitute study medication for their pre study prescribed asthma medication for the duration of the study.
* Written informed parental consent obtained, and where possible informed assent from the patient.

Exclusion Criteria:

* Life-threatening asthma within the past year. This category includes those patients with a history of near-fatal asthma, a hospitalization or an emergency visit for asthma or prior intubation for asthma.
* History of systemic (injectable) corticosteroid medication within 1 month before the Screening Visit.
* History of leukotriene receptor antagonist use, e.g. montelukast, within the past week.
* Current evidence or history of any clinically significant disease or abnormality including uncontrolled coronary artery disease, congestive heart failure, or cardiac dysrhythmia. 'Clinically significant' is defined as any disease that, in the opinion of the Investigator, would put the patient at risk through study participation, or which would affect the outcome of the study.
* An upper or lower respiratory infection within 4 weeks prior to the Screening Visit.
* Significant, non-reversible, active pulmonary disease (e.g., chronic obstructive pulmonary disease (COPD), cystic fibrosis, bronchiectasis, tuberculosis).
* Known Human Immunodeficiency Virus (HIV)-positive status.
* Current smoking history within 12 months prior to the Screening Visit.
* Current evidence or history of alcohol and/or substance abuse within 12 months prior to the Screening Visit.
* Patients who have taken B-blocking agents, tricyclic antidepressants, monoamine oxidase inhibitors, astemizole (Hismanal), quinidine type antiarrhythmics, or potent CYP 3A4 inhibitors such as ketoconazole within the past week.
* Current use of medications that will have an effect on bronchospasm and/or pulmonary function.
* Current evidence or history of hypersensitivity or idiosyncratic reaction to test medications or components.
* Receipt of an investigational drug within 30 days of the Screening Visit (12 weeks if an oral or injectable steroid).
* Current participation in a clinical study.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 211 (Actual)
Dates: Start 2007-03; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
FEV1, recorded at visits to investigator at 2 wks, 6wks & 12 wks.

SECONDARY OUTCOMES:
Lung function tests, peak expiratory flow rate, asthma symptoms & exacerbations, adverse events, sleep disturbance, rescue medication use, plasma cortisol (extension only).

CONTACTS AND LOCATIONS:
Locations (6):
- Prague, Czechia
- Laon, France
- Wiesal, Germany
- Budapest, Hungary
- Lublin 20-093, W. Chodzki 2, Poland
- Bucharest, Romania

REFERENCES:
- See also: Results available on website — https://www.clinicaltrialsregister.eu/ctr-search/search?query=FLT3502